CLINICAL TRIAL: NCT04362943
Title: Clinical-epidemiological Characterization of COVID-19 Disease in Hospitalized Older Adults
Acronym: COVID-AGE
Status: Completed | Type: Observational
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Responsible Party: Principal Investigator, Pedro Abizanda, Prof., Complejo Hospitalario Universitario de Albacete
Other Study IDs: PAS-BAR-2020-04
Record Dates: First submitted 2020-04-22; First posted 2020-04-27 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
Keywords: COVID-19; Older adults; Hospitalization; Baricitinib; Anakinra; Effectiveness; Security; Mortality
MeSH Terms: conditions — COVID-19 | interventions — baricitinib; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Complete sample: Adults older than 70 years hospitalized for COVID-19 disease between 09/03/2020 and 20/04/2020 in the "Perpetuo Socorro" Hospital of Albacete (Spain)
  Interventions: Drug: Baricitinib or Anakinra
- Baricitinib: Adults older than 70 years hospitalized for COVID-19 disease between 09/03/2020 and 20/04/2020 and receiving Baricitinib.
  Interventions: Drug: Baricitinib or Anakinra
- Anakinra: Adults older than 70 years hospitalized for COVID-19 disease between 09/03/2020 and 20/04/2020 and receiving Anakinra.
  Interventions: Drug: Baricitinib or Anakinra

INTERVENTIONS:
Drug: Baricitinib or Anakinra — Treatment with either Baricitinib or Anakinra during hospitalization, in real world, and under usual clinical care.

SUMMARY:
Retrospective clinical-epidemiological study aimed at characterizing COVID-19 disease in adults older than 70 years, hospitalized in the "Perpetuo Socorro" Hospital of Albacete (Spain) from 09/03/2020 until 20/04/2020. Secondary objectives will be to analyze clinical-epidemiological characteristics of COVID-19 patients treated with Baricitinib or Anakinra, and to describe the efficacy and secondary effects of those drugs.

DETAILED DESCRIPTION:
Design: Retrospective postauthorization study. Registry study. Setting: COVID Unit, "Perpetuo Socorro" Hospital of Albacete (Spain). Participants: Adults older than 70 years hospitalized for COVID-19 disease between 09/03/2020 and 20/04/2020. All patients will be included without exclussion criteria.

Measurements:

* Age, sex, residency.
* Functional assessment: Barthel index, Katz index, Functional Ambulation Classification.
* Cognitive assessment: Reisberg´s Global Deteriorating Scale.
* Comorbidity: Charlson index, disease count.
* Chronic medicines consumed.
* Disease related symptoms.
* Lab determinations: White cells, neutrophyl count, lymphocyte count, platelets, haemoglobin, INR, fibrinogen, D-Dimer, Ferritin, CRP, IL-6, urea, creatinin, AST, ALT, CK.
* Thorax X-ray findings: COVID affectation, severity, pleural effusion, heart failure signs, pneumothorax.
* Drugs used during hospitalization, number of days of treatment and total doses: Anakinra, Baricitinib, Glucocorticoids, Antivirals (Lopinavir/Ritonavir, Emtricitabina/Tenofovir), Azitromycin, Ceftriaxone, Hidroxychloroquin.
* Geriatric syndroms: Delirium, immobility, dysphagia, pressure ulcers.
* Outcomes: Mortality at discharge, institucionalización at discharge, length of stay, change in lab results, change in X-ray results, change in function at discharge.

Registry procedures: Medical chart review by trained Geriatricians, pharmachological chart review by expert Pharmacists, X-ray review by trained radiologists. All data will be included in an anonimyzed database for further analysis by investigators, and supervised by Principal Investigator.

Regulatory status: The protocol was approved by the Ethics review committee of Albacete (number 2020-21 from 20/04/2020) and by the Spanish Medicines Agency (AEMPS) who gave a "Postauthorization Study" classification (number PAS-BAR-2020-04. 20/04/2020).

Analysis: Two stage analysis will be conducted. In first one, efficacy and security analysis of the 99 patients that have received either Baricitinib or Anakinra will be conducted, and in the second one, clinical-epidemiological analysis of the complete sample, n=576, will be realized.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 70 years hospitalized for COVID-19 disease between 09/03/2020 and 20/04/2020, in the "Perpetuo Socorro" Hospital of Albacete (Spain).

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults older than 70 years hospitalized for COVID-19 disease between 09/03/2020 and 20/04/2020, in the "Perpetuo Socorro" Hospital of Albacete (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 month
  Mortality for all causes

SECONDARY OUTCOMES:
X-ray changes | 1 month
  Changes from admission to discharge thorax X-rays assessed by blinded radiologists
Disability changes | 1 month
  Changes from admission to discharge in Barthel index
Ambulation changes | 1 month
  Changes from admission to discharge in Functional Ambulation Classification
lymphocyte count changes | 1 month
  Changes from admission to discharge in lymphocyte count
C-Reactive Protein changes | 1 month
  Changes from admission to discharge in C-Reactive Protein
Ferritin changes | 1 month
  Changes from admission to discharge in Ferritin
D-Dimer changes | 1 month
  Changes from admission to discharge in D-Dimer

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Abizanda Soler, MD,PhD, Principal Investigator — Head Geriatrics Department
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request. Study protocol, statistical analysis and clinical study report will be shared when data will be published in a Journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At data Journal publication